Study Title: Efficacy of a Dissonance Based Eating Disorder Program

NCT Number: 03796091 ID: 1516-105-GRE

Date of IRB Approval: May 8, 2018 (updated analysis plan approved)

Document Type: Analysis Plan
Pl: Dr. Melinda Ann Green
Institution: Cornell College

Eating disorder symptoms, body dissatisfaction, negative affect, positive affect, state anxiety, thin-ideal internalization, maladaptive social comparison, self-objectification, mean R wave amplitude, QT interval length, sympathetic tone (LF/HF spectral power ratio), and HF power will be evaluated at baseline, postintervention, and 2-month follow-up. Single mean imputation will be used to impute missing values so that all statistical tests will be conducted on the complete dataset (N=180) with missing values imputed. We predict a statistically significant 3 (group: enhanced dissonance, traditional dissonance, educational brochure control) x 3 (time: baseline, postintervention, 2-month follow-up) interaction in mixed factorial MANOVA results. Specifically, we predict participants in the enhanced dissonance condition will show lower levels of eating disorder symptoms and associated risk factors compared to participants in the control or traditional dissonance conditions at postintervention and 2-month follow-up as indicated by follow up tests including a series of 3 (group) x 3 (time) ANOVAs and posthoc comparisons for each dependent variable. The data analysis strategy outlined above assumes data meet normality (skewness and kurtosis) assumptions. If these assumptions are not met, the PI will consult with the Cornell College Quantitative Reasoning Studio Consultant to assist with conducting the relevant non-parametric tests.